CLINICAL TRIAL: NCT02346864
Title: Effect of Three-Stair-Position on Improvement of Apnea of Prematurity and Feeding Performance in Prematurity: A Randomized Control Trial
Brief Title: Effect of Three-Stair-Position on Improvement of Apnea of Prematurity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: FNF201221
Record Dates: First submitted 2014-12-25; First posted 2015-01-27 (Estimated); Last update posted 2015-01-27 (Estimated); Status verified 2015-01

CONDITIONS: Apnea of Prematurity
Keywords: head elevated position; preterm; three-stair-position
MeSH Terms: conditions — Apnea; Premature Birth

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Three-stair-position group (Experimental): The infants in the study group (n=72) received three-stair-position (TSP) intervention (head up 15°) for a week.
  Interventions: Behavioral: Three-stair-position
- head elevated tilt position group (Other): The control group(n=72)received head elevated tilt position (HETP) intervention (head up 15°) for a week．
  Interventions: Behavioral: Head elevated tilt position group

INTERVENTIONS:
Behavioral: Three-stair-position — Infants in the TSP group received three-stair-prone position. Implementation steps were as following: 1) produced pad of three-stair-prone position the total height of which should be the same height as the head elevated 15 °. 2) Placed the infants on the pad with head on the highest ladder, chest on the second step and leg on the third step, bending the knees to the chest
  Arms: Three-stair-position group
Behavioral: Head elevated tilt position group — Infants in the HETP group were allowed head up 15 ° prone position using a protractor with head to one side, arms against the sides of the body naturally bending, knees bent to the chest.
  Arms: head elevated tilt position group

SUMMARY:
The purpose of this study is evaluating the effectiveness of three-stair-position (TSP) on the rate of Apnea of Prematurity (AOP), the feeding performance and the vital signs.

DETAILED DESCRIPTION:
Apnea of Prematurity (AOP) is common critical symptoms of preterm infants with great harm for prematurity. Recurrent apnea may lead to brain damage caused by hypoxia, affecting the nervous system, even threatening life (1, 2). Therefore, choosing an intervention which can prevent and reduce occurrence of AOP with fewer side effects is an important issue that should be closely watched by neonatal intensive care unit (NICU) health care.

Prone position is the forefront treatment due to its simple, economic and non-invasive. In clinic, it includes horizontal prone position (HPP), Head elevated tilt 15 ° prone position (HETP) and three-step-prone position (TSP)(3).Many studies have shown that HETP can allow thoracic volume increased and make abdominal movement more coordinated in preterm children, and then it is more favorable than the HPP on improving respiratory function. So HETP has been a routine position in NICU instead of HPP (4, 5). HETP, however, always make the babies slide to the foot of the bed resulting in airway obstruction. Therefore, scholars have proposed TSP which should prevent this phenomenon (6). In the study, the effectiveness of TSP on improvement of AOP will be evaluated trying to find a more suitable position for preterm infants.

ELIGIBILITY:
Inclusion Criteria:

1. preterm, gestational age(GA) <34weeks determined by obstetric ultra-sonogram and clinical examination
2. steady vital signs
3. Apgar scores were greater than or equal to 3 at 1min and greater than or equal to 5 at 5 minutes.

Exclusion Criteria:

1. infants with congenital malformation，for example Congenital Heart Disease, Diaphragmatic hernia, Hirschsprung,etc
2. Infants who need special position and/or intervention (gastroschisis or umbilical catheterization)
3. weight<1000g
4. infants who were undertaking conventional invasive mechanical ventilation.

Max Age: 3 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 144 (Actual)
Dates: Start 2013-12; Primary Completion 2014-08 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
The rate of AOP | 7 Days
Frequency of desaturation which defined as oxygen saturation by pulse oximetry (SPO2)<85% | 7 Days

SECONDARY OUTCOMES:
Number of Participants who need treatments | 7 Days
  Treatments of AOP include stimulation, nasal cannula oxygen, pressurized oxygen, continuous positive airway pressure (CPAP), invasive mechanical ventilation, medication (pulmonary surfactant, aminophylline).
Adverse events during feeding | 7 Days
Times of milk retention | 7 Days
Number of Participants with distension | 7 Days
  Distension was diagnosed by a doctor and a nurse.
Heart rate | 7 Days
Number of Participants with Adverse Events | 7 Days
amount of retention milk | 7 Days
respiratory rate | 7 Days
SPO2 | 7 Days